CLINICAL TRIAL: NCT03405649
Title: Active Mother- Active Baby: Resistance Training in Postpartum Women as a Group Class Exercise Intervention With Their Babies.
Brief Title: Active Mother May Lead to an Active Baby.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Michelle Mottola, Professor, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110303
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Postpartum; Exercise; Intervention
Keywords: postpartum; exercise; intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Women contacting the lab will be divided into those women who have babies less than 20 weeks of age (Group A) and those whose babies are greater than 20 weeks of age (Group B). Each of these groups will be given a separate postpartum exercise program that will run concurrently. These groups were divided by baby age because we felt early postpartum women and babies are a different group than those women with babies 6 months and older.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants train 60 min per session for 10 weeks on non-consecutive days. All training sessions will be supervised by a qualified exercise instructor. Each training session will include a warm up phase of 5 minutes of dynamic and static stretching and a cool down phase consisting of 5 minutes of static stretching. Whole-body exercises and weights, elastic bands and balls will be used. Babies less than 20 weeks of age will be included in the exercise routine. Participants will perform 1-3 sets per exercise, 8-12 repetitions per set and a 90-s rest interval between sets.
  Interventions: Behavioral: Group A
- Group B (Experimental): Participants train 60 min per session for 10 weeks on non consecutive days. All training sessions will be supervised by a qualified exercise instructor. Each training session will include a warm up phase of 5 minutes of dynamic and static stretching and a cool down phase consisting of 5 minutes of static stretching. Whole-body exercises and different equipment such as weights, elastic bands and balls will be used. Babies older than 20 weeks will be included in the exercise routine. Participants will perform 1-3 sets per exercise, 8-12 repetitions per set and a 90-s rest interval between sets.
  Interventions: Behavioral: Group B

INTERVENTIONS:
Behavioral: Group A — Muscle conditioning exercise for postpartum women and infants less than 20 weeks of age.
  Arms: Group A
Behavioral: Group B — Muscle conditioning exercise for postpartum women and infants more than 20 weeks of age.
  Arms: Group B

SUMMARY:
Among the well-known factors that contribute to the development of obesity, childbearing has been reported as an important influential factor. Physical activity is strongly recommended as one of the main tools to reduce any excessive weight gain during pregnancy and also to reduce weight retention in the postpartum period. During the postpartum period, exercise training coupled with a well-balanced nutritional plan, offers an effective intervention to help mothers lose weight safely. International guidelines for physical activity after pregnancy include strengthening routines. Worth noting, most of the above cited studies focused on the benefits of aerobic activities. Strength training interventions are virtually unexplored in postpartum women despite its potential benefits. Compared to the pregnancy period, postpartum barriers to physical activity seem to focus less on health-related barriers. In postpartum, time limitations for childcare become a more common barrier. For this reason, a postpartum exercise program that incorporates the babies in a specific exercise session has a better chance to succeed. The aim of this project is to determine the benefits of strength training in a group class setting in postpartum healthy women with their babies. Whereas mother's participation in regular physical activity may encourage regular physical activity habits in her offspring, a second aim of this project is to also quantify the infant's physical activity. The main measured outcomes are: maternal muscular strength; body composition; aerobic capacity; exercise self efficacy; depressive symptoms; physical activity level and food habits and baby's physical activity level.

DETAILED DESCRIPTION:
Research Questions:

Maternal:

Is a strength training group class (with babies) in postpartum women associated with (I) strength and lean body mass improvement, (II) improvement aerobic capacity, (III) more spontaneous physical activity, (IV) better self efficacy and (V) better mood?

Baby:

Does maternal lifestyle affect the baby's (0-12 months) physical activity level?

Hypothesis:

It is hypothesized that women who complete the 10 week exercise program will have improved strength from pre-intervention to post intervention. It is also hypothesized that women who are adherent to the exercise program will have more active babies.

Methods:

Participants train 60 min per session for 10 weeks on non consecutive days (Tues and Thurs). All training sessions will be supervised by a qualified exercise instructor (graduate in kinesiology) to ensure proper technique and to minimize the risk of injury. Each training session will include a warm up phase of 5 minutes of dynamic and static stretching and a cool down phase consisting of 5 minutes of static stretching. The strength training protocol is based on the American College of Sports Medicine (ACSM) guidelines. Whole-body exercises and different equipment such as weights, elastic bands and balls will be used. Babies will also be included in the exercise routine. Participants will perform 1-3 sets per exercise, 8-12 repetitions per set and a 90-s rest interval between sets. The principle of progressive overload will follow a linear increase as described in ACSM position stand.

All participants will be tested at time points t0 , t1 ( after 5 weeks) and t2 (after 10 weeks; at the and of the study) on: i) strength and body composition; ii) aerobic capacity; iii) objective and subjective physical activity level; vi) exercise self efficacy; v) depressive symptoms and vi) dietary habits.

I. Strength/Body composition assessment At each time point, strength will be assessed for the upper body (push-ups), lower body (squats), and trunk (abdominal curl-up test). The participants will perform push-ups (as many as possible using a fixed pattern of 40 beats per minute - time and number will be recorded up to a maximum of 1 minute). This will be repeated for the number of lower body squat position performed (as many squats as possible using a fixed pattern of 40 beats per minute -time and number will be recorded up to a maximum of 1 minute); these methods have been chosen to reduce the likelihood of any adverse events. The participant will also complete the ACSM-recommended partial curl-up test to assess abdominal strength and endurance. Briefly, as many abdominal curl-ups as possible has to be performed until the participant either stops, or cannot stay in rhythm with a fixed cadence (40 beats/min) up to 1 minute as per ACSM guidelines.

Body composition assessment will include body mass, height, BMI and body fat (sum of five skinfolds: triceps, biceps, subscapular, suprailiac, thigh) measures.

II. Aerobic capacity Briefly, participants perform a 5- min. bout of exercise, stepping up and down from a standard step (height 30 cm) following a specific cadence. During the step test, heart rate (HR) is measured continuously using a heart-rate monitor. Then, VO2max is estimated based on HR and a target exercise intensity (estimated VO2).

III. Physical activity assessment At each time point, participants will to complete two self- reported questionnaires regarding physical activity level, the International Physical Activity Questionnaire (IPAQ; and the Physical Activity Readiness Questionnaire (PAR-Q+).The IPAQ asks participants to recall their levels of physical activity within five domains (leisure, work, transportation, household, recreation) and three intensity categories over a 7-day recall period. The PAR-Q+ determines if it is safe to start an exercise program. Additionally, at t0, t1 and t2 each participant will complete an individual physical activity diary for 7 days. Moreover, during this period participants will continuously wear a pedometer .

IV. Exercise self efficacy Exercise self-efficacy will be measured at each time point (t0,t1 and t2). This survey includes five separate items targeting self-efficacy.

V. Depressive symptoms Levels of postpartum mood will be assessed through the Edinburgh Postnatal Depression Scale (EPDS).

VI. Eating Habits Mother's eating habits will be measured through the Short-Form Frequency Questionnaire (SFFFQ).

VII. Breastfeeding habits will be measured through a Breastfeeding and Infant Feeding Questionnaire.

Baby At each time point, a Rothbart Infant Behavior Questionnaire- Revised (IBQ-R) will be completed by the participants to measure temperament and gross motor activity in infants between the ages of 3 and 12 months.

This study will take place at the Canadian Centre for Activity and Aging gymnasium on Tuesday and Thursday afternoons (time to be determined). Women who contact us will be asked when their baby was born. Those women whose babies are less than 20 weeks of age will be placed in Group A and those women whose babies are older than 20 weeks will be placed in Group B. These groups were divided by baby age because early postpartum women and babies are a different group than those women with babies 6 months and older.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (free from chronic diseases) women between 8 weeks and 50 weeks after delivery.

Exclusion Criteria:

* Inability to perform strength training or moderate-intensity exercise, athletes/well trained mothers (i.e. mothers undergoing regular strength training), smokers and women who are planning to become pregnant over the subsequent year. Women who cannot read, write and understand English will not be included.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postpartum women and their infants of both sexes.
Enrollment: 60 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Maternal overall muscular strength | 10 weeks
  A series of muscular strength assessments will be performed at baseline, after 5 weeks and at 10 weeks of intervention. Higher number of timed push-ups, squats and sit-ups increased from baseline will indicate improved muscular strength.

SECONDARY OUTCOMES:
Maternal body composition | 10 weeks
  Maternal skinfolds will be assessed at baseline, after 5 weeks and at 10 weeks of intervention. Decreased skinfold measurements from baseline will indicate improved body composition and loss of body fat.
Maternal aerobic capacity | 10 weeks
  Maternal oxygen consumption will be measured at baseline, after 5 weeks and at 10 weeks of intervention. Improvement in aerobic capacity will be indicated by higher estimated VO2 measurements at the end of the intervention compared to baseline.
Maternal physical activity level measured by the International Physical Activity Questionnaire (IPAQ) | 10 weeks
  Using the IPAQ, physical activity will be measured at baseline, after 5 weeks and at 10 weeks of intervention. Based on the IPAQ vigorous activity is 8 METmin/day; moderate activity is 4 METmin/day and light activity is 3 METmin/day. Total activity will be the addition of vigorous, moderate and light activities recorded in METmin/day. Total METmin/day that is <700 is defined as "inactive"; 700-2519 METmin/day is defined as "active" and > 2520 METmin/day is defined as "very active". An increase in physical activity will be indicated by an increase in total METmin/day from baseline to end of intervention.
Maternal self-efficacy | 10 weeks
  Women will complete a self-efficacy questionnaire at baseline, after 5 weeks and at 10 weeks at the end of the intervention. Improvement in self-efficacy will be indicated by an increase in total score from baseline.
Maternal eating habits | 10 weeks
  Women will complete a food frequency questionnaire at baseline, after 5 weeks and at 10 weeks at the end of the intervention. Dietary habits will be improved from baseline if women eat more healthy foods such as vegetables and fruit and decrease intake of high density foods such as junk food.
Maternal breast feeding behavior | 10 weeks
  Women will complete a breast feeding questionnaire at baseline, after 5 weeks and at 10 weeks at the end of the intervention. This questionnaire includes frequency of breast feeding and whether infant feeding is supplemented by formula. This is self-reported and descriptive to describe breast feeding behavior.
Gross motor activity using the Rothbart Infant Behavior Questionnaire- Revised (IBQ-R) | 10 weeks
  Women will complete only the activity component of the Rothbart Infant Behavior Questionnaire- Revised (IBQ-R) that contains 15 items to assess infant gross motor activity at baseline, after 5 weeks and at 10 weeks at the end of the intervention. Each question is answered using a 7 point scale (indicating activity over the last 7 days). The scare ranges from 1 - "never", 2 - "very rarely", 3 - "< half the time", 4 - "about half the time", 5 - "> half the time", 6 - "almost always", 7 - "always". The score for the 15 questions is totaled. The higher the score, the more active the infant in gross motor activity. A perfect score is 105 and at each time point the total activity scores will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Mottola, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- Exercise and Pregnancy Lab, 2245, 3-M Centre - University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available within 1 year of study completion.
Access Criteria: Data access requests will be reviewed by an independent review panel. Requestors will be required to sign a data access agreement and privacy statement.